CLINICAL TRIAL: NCT06972862
Title: Optimizing Muscle and Bone Mechanoadaptation to Physical Training: Mechanistic Control Paths Via Muscle and Bone Crosstalk to Altered Mechanical Loading
Brief Title: Bone and Body Composition Adaptations to Physical Training
Acronym: BoBCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Bradley Nindl, Professor and Vice Chair for Research, Department of Sports Medicine and Nutrition, University of Pittsburgh; Director, Neuromuscular Research Laboratory/Warrior Human Performance Research Center, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21020044; W81XWH-21-1-0542 (Other Grant/Funding Number: Department of Defense, USAMRAA)
Record Dates: First submitted 2025-04-28; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Exercise; Healthy
Keywords: bone health; body composition; skeletal muscle; hormones; exercise intervention; recreational athletes; bone marrow adipose tissue; bone formation; bone resportion; bone geometry; bone microarchitecture; bone mineral density
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laboratory Based Osteogenic Index (OI) Optimized Training Group (Experimental): The OI- Optimized Training Group will involve 6 months of planned, non-linear periodized training on a leg press machine called the PPM (Athletic Republic, Salt Lake City, UT) with a maintenance program during the semester breaks, as necessary.
  Interventions: Other: Osteogenic Index Optimized Exercise Training Program
- Laboratory Based Control Group (No Intervention): The control group will maintain their habitual exercise, diet, and sleep patterns, all of which will be monitored throughout the study.
- Reserve Officer Training Corps (ROTC): Observational Group (No Intervention): The ROTC group is made up of Reserve Officer Training Corps participants who are attending a university while concurrently undergoing militaristic training. This group will maintain their physical training as part of their program, diet, and sleep patterns which are monitored throughout the study.

INTERVENTIONS:
Other: Osteogenic Index Optimized Exercise Training Program — The OI- Optimized Training is 6 months of planned, non-linear periodized training on a leg press machine called the PPM (Athletic Republic, Salt Lake City, UT) with a maintenance program during the semester breaks, as necessary.
  Other Names: Exercise Intervention
  Arms: Laboratory Based Osteogenic Index (OI) Optimized Training Group

SUMMARY:
The goal of this clinical trial is to evaluate how different exercise programs alter bone density, structure, and strength in adults. It will also collect data on hormones, factors released from skeletal muscle, and body composition.

The main questions it aims to answer are:

* Do exercise programs that are frequent with high-impact loading will cause greater improvements in bone health?
* What changes in hormones, factors released from skeletal muscle, and body composition contribute to bone adaptations?

Researchers will compare different exercise groups to see if the type of exercise influences bone adaptation compared to a recreationally active control group.

Participants are asked to:

* complete questionnaires, 5 blood draws across the study (3 at rest, 2 after strenuous exercise), dual energy x-ray absorptiometry (DXA) scans (to assess bone mineral density and body composition), high resolution tibial scans to assess bone structure and geometry, and physical performance testing.
* attend up to 7 testing visits.
* (for those randomized to the exercise training intervention) participate in exercise training sessions for 6 months.

DETAILED DESCRIPTION:
The overall objective of this study is to determine the bone density, structure and strength adaptations that result from various exercise programs which differ based on the frequency and intensity of bone loading. Bone adaptation is measured with both dual-energy x-ray absorptiometry (DXA), the standard-of-care equipment used to evaluate bone mineral density (BMD), and high-resolution peripheral quantitative computed tomography (HRpQCT), a state-of-the-science imaging technology providing the resolution necessary to detect small but clinically relevant changes.

Additionally, the research team seeks to determine the physiological responses and adaptations to training that contribute to improved bone health by evaluating changes in hormones, factors released from active skeletal muscle, and body composition. Our hypothesis is that exercise programs emphasizing frequent, high impact loading will cause greater improvements in bone health. Additionally, we believe that exercise training can induce specific changes in hormones, skeletal muscle released signaling factors and body composition that contribute to these bone adaptations.

Participants who enrolled in this study were randomized to either an exercise training group or a control group who were instructed to maintain their current level of exercise and track this to report to the study team. Study completers were those who complied with the parameters of the group they were assigned and reported to all 7 testing visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-40 years
2. Body mass index (BMI) 18-28 kg/m2
3. Weight stable (±10 lbs) in past 2 months
4. Takes part in moderate physical activity for at least 150 minutes/week
5. Currently free of upper or lower body /extremity injury or impairment
6. Comfortable with multiple blood draws
7. Able to commit to the 6-month study duration
8. Agrees to adhere to study requirements.

Exclusion Criteria:

1. Current smoker
2. Current clinical diagnosis of an eating disorder
3. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs). NSAID use is defined as chronic if these medications are taken more than three times a week for more than 12 consecutive weeks.
4. Use of medication incompatible with measurement of reproductive, metabolic, or bone-related hormones (including thyroid medications, glucocorticoids) or which includes anti-coagulants and may interfere with any of the study outcomes
5. Current oligo/amenorrhea in women, not explained by contraceptive use
6. Any metabolic or endocrine disease that affects bone; Individuals taking hormonal therapy for transgender care
7. Currently training for a competitive sporting event or planning to start
8. Weight has fluctuated by 10 pounds or more in the past 2 months based on subject self-report
9. Has been diagnosed with a medical condition, physical or psychological, that currently prevents exercise participation
10. Has suffered a musculoskeletal injury removing them from physical activity for more than a month, within the past two years
11. Currently pregnant or becomes pregnant during the study (as assessed by urine pregnancy tests at 0, 3 & 6 months)
12. Current asthma diagnosis, defined as experienced symptoms or been prescribed any form of treatment within the last 4 years, or those who have required more than one course of oral steroids or more than one nebulization since the age of 5 (JSP 950), will require a note/permission from treating physician to participate in study. Those who have had a single admission to intensive care or high dependency, or multiple admissions to hospital will be excluded from participating (JSP 950)
13. History of heart condition OR high blood pressure
14. Feeling of pain in the chest during rest, activities of daily living, or physical activity
15. Have lost balance or consciousness due to dizziness in the last 12 months (with the exception of dizziness due to hyperventilation)
16. Treating physician requires subject participates in medically supervised physical activity only
17. History of drug addiction or habitual recreational drug use (2 or more times per month in each of the previous six months)
18. Low bone mineral density indicated as a Z-score <-1.0 measured by dual-energy x-ray absorptiometry (DXA)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 206 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2025-04-27 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Bone microarchitecture: Change in bone microarchitecture as measured via High Resolution- peripheral Quantitative Computed Tomography, change from baseline, mean | Through study completion, an average of 6 months.
Bone strength: Change in bone strength as measured via High Resolution- peripheral Quantitative Computed Tomography, change from baseline, mean | Through study completion, an average of 6 months

SECONDARY OUTCOMES:
Biochemical: Change in concentration of Bone alkaline phosphatase (BAP), change from baseline, mean | Through study completion, an average of 6 months
  BAP is a bone formation marker.
Biochemical: Change in concentration of Procollagen type I N-terminal Propeptide (P1NP), change from baseline, mean | Through study completion, an average of 6 months
  P1NP is a bone formation marker.
Biochemical: Change in concentration of Tartrate-resistant acid phosphatase 5b (TRAP5b), change from baseline, mean | Through study completion, an average of 6 months
  TRAP5b is a bone resorption marker.
Biochemical: Change in concentration of Beta Cross-linking Telopeptide of type I (B-CTx) collagen, change form baseline, mean | Through study completion, an average of 6 months
  B-CTx is a bone resorption marker.
Bone characteristics: Change in amount of Bone Marrow Adipose Tissue, change from baseline, mean | Through study completion, an average of 6 months
Biochemical: Change in extracellular vesicle size, change from baseline and through study completion, mean | Through study completion, an average of 6 months
  This is a descriptive analysis in which the mean size of the extracellular vesicles will be assessed via nanoparticle tracking analysis between groups and throughout the study.
Biochemical: Change in extracellular vesicle constituent cargo, change from baseline and through study, mean | Through study completion, an average of 6 months
  This is a descriptive analysis in which the mean contents of the extracellular vesicles will be assessed via proteomics between groups and throughout the study.
Biocehmical: Rate of change in micro- RNA expression, from baseline through study completion, Log2 Fold Change between groups | Through study completion, an average of 6 months
  A descriptive analysis will be performed in which the micro-RNA expression in each group will be compared via the Log2 Fold Change (a type of rate of change) mathematical formula (Log2 Fold Change (LogFC): log2(Expression Level (Group 1) / Expression Level (Group 2))).

OTHER OUTCOMES:
Body composition: Change in Dual Energy X-Ray Absorptiometry lean mass, change from baseline, mean | Through study completion, an average of 6 months
Bone characteristics: Change in Areal Bone Mineral Density, change from baseline, mean | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristen J Koltun, PhD, Study Director — University of Pittsburgh
Locations (2):
- United States (2):
  - University of Kansas, Jayhawk Performance Laboratory, Lawrence, Kansas
  - Neuromuscular Research Laboratory, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after identification (text, tables, figures, and appendices).
Time Frame: Beginning 1 year and ending 5 years following publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. For individual participant data meta-analysis. Proposals should be directed to bnindl@pitt.edu. To gain access, data requesters will need to sign a data access agreement.

REFERENCES:
- [Background] Allaway HC, Williams NI, Mallinson RJ, Koehler K, De Souza MJ. Reductions in urinary collection frequency for assessment of reproductive hormones provide physiologically representative exposure and mean concentrations when compared with daily collection. Am J Hum Biol. 2015 May-Jun;27(3):358-71. doi: 10.1002/ajhb.22649. Epub 2014 Oct 29. PMID 25353669
- [Background] Nindl BC, Urso ML, Pierce JR, Scofield DE, Barnes BR, Kraemer WJ, Anderson JM, Maresh CM, Beasley KN, Zambraski EJ. IGF-I measurement across blood, interstitial fluid, and muscle biocompartments following explosive, high-power exercise. Am J Physiol Regul Integr Comp Physiol. 2012 Nov 15;303(10):R1080-9. doi: 10.1152/ajpregu.00275.2012. Epub 2012 Aug 29. PMID 22933025
- [Background] Lester ME, Urso ML, Evans RK, Pierce JR, Spiering BA, Maresh CM, Hatfield DL, Kraemer WJ, Nindl BC. Influence of exercise mode and osteogenic index on bone biomarker responses during short-term physical training. Bone. 2009 Oct;45(4):768-76. doi: 10.1016/j.bone.2009.06.001. Epub 2009 Jun 9. PMID 19520194
- [Background] Carson JA, Manolagas SC. Effects of sex steroids on bones and muscles: Similarities, parallels, and putative interactions in health and disease. Bone. 2015 Nov;80:67-78. doi: 10.1016/j.bone.2015.04.015. PMID 26453497
- [Background] Wentz L, Liu PY, Haymes E, Ilich JZ. Females have a greater incidence of stress fractures than males in both military and athletic populations: a systemic review. Mil Med. 2011 Apr;176(4):420-30. doi: 10.7205/milmed-d-10-00322. PMID 21539165
- [Background] Rantalainen T, Nikander R, Heinonen A, Cervinka T, Sievanen H, Daly RM. Differential effects of exercise on tibial shaft marrow density in young female athletes. J Clin Endocrinol Metab. 2013 May;98(5):2037-44. doi: 10.1210/jc.2012-3748. Epub 2013 Apr 24. PMID 23616150
- [Background] Singhal V, Torre Flores LP, Stanford FC, Toth AT, Carmine B, Misra M, Bredella MA. Differential associations between appendicular and axial marrow adipose tissue with bone microarchitecture in adolescents and young adults with obesity. Bone. 2018 Nov;116:203-206. doi: 10.1016/j.bone.2018.08.009. Epub 2018 Aug 11. PMID 30107255
- [Background] Gorgey AS, Poarch HJ, Adler RA, Khalil RE, Gater DR. Femoral bone marrow adiposity and cortical bone cross-sectional areas in men with motor complete spinal cord injury. PM R. 2013 Nov;5(11):939-48. doi: 10.1016/j.pmrj.2013.05.006. Epub 2013 May 15. PMID 23684921
- [Background] Sanford JA, Nogiec CD, Lindholm ME, Adkins JN, Amar D, Dasari S, Drugan JK, Fernandez FM, Radom-Aizik S, Schenk S, Snyder MP, Tracy RP, Vanderboom P, Trappe S, Walsh MJ; Molecular Transducers of Physical Activity Consortium. Molecular Transducers of Physical Activity Consortium (MoTrPAC): Mapping the Dynamic Responses to Exercise. Cell. 2020 Jun 25;181(7):1464-1474. doi: 10.1016/j.cell.2020.06.004. PMID 32589957
- [Background] Whitham M, Parker BL, Friedrichsen M, Hingst JR, Hjorth M, Hughes WE, Egan CL, Cron L, Watt KI, Kuchel RP, Jayasooriah N, Estevez E, Petzold T, Suter CM, Gregorevic P, Kiens B, Richter EA, James DE, Wojtaszewski JFP, Febbraio MA. Extracellular Vesicles Provide a Means for Tissue Crosstalk during Exercise. Cell Metab. 2018 Jan 9;27(1):237-251.e4. doi: 10.1016/j.cmet.2017.12.001. PMID 29320704
- [Background] Norheim F, Langleite TM, Hjorth M, Holen T, Kielland A, Stadheim HK, Gulseth HL, Birkeland KI, Jensen J, Drevon CA. The effects of acute and chronic exercise on PGC-1alpha, irisin and browning of subcutaneous adipose tissue in humans. FEBS J. 2014 Feb;281(3):739-49. doi: 10.1111/febs.12619. Epub 2013 Dec 10. PMID 24237962
- [Background] Robling AG, Niziolek PJ, Baldridge LA, Condon KW, Allen MR, Alam I, Mantila SM, Gluhak-Heinrich J, Bellido TM, Harris SE, Turner CH. Mechanical stimulation of bone in vivo reduces osteocyte expression of Sost/sclerostin. J Biol Chem. 2008 Feb 29;283(9):5866-75. doi: 10.1074/jbc.M705092200. Epub 2007 Dec 17. PMID 18089564
- [Background] Bonewald LF, Johnson ML. Osteocytes, mechanosensing and Wnt signaling. Bone. 2008 Apr;42(4):606-15. doi: 10.1016/j.bone.2007.12.224. Epub 2008 Jan 12. PMID 18280232
- [Background] Evans RK, Negus CH, Centi AJ, Spiering BA, Kraemer WJ, Nindl BC. Peripheral QCT sector analysis reveals early exercise-induced increases in tibial bone mineral density. J Musculoskelet Neuronal Interact. 2012 Sep;12(3):155-64. PMID 22947547
- [Background] Hughes JM, Gaffney-Stomberg E, Guerriere KI, Taylor KM, Popp KL, Xu C, Unnikrishnan G, Staab JS, Matheny RW Jr, McClung JP, Reifman J, Bouxsein ML. Changes in tibial bone microarchitecture in female recruits in response to 8 weeks of U.S. Army Basic Combat Training. Bone. 2018 Aug;113:9-16. doi: 10.1016/j.bone.2018.04.021. Epub 2018 Apr 27. PMID 29709620
- See also: Neuromuscular Research Laboratory Website — https://www.nmrl.pitt.edu

DOCUMENTS (1):
  • Informed Consent Form (2024-04-16): https://cdn.clinicaltrials.gov/large-docs/62/NCT06972862/ICF_000.pdf